CLINICAL TRIAL: NCT03066271
Title: PRIME - Pre Radiotherapy Daily Exercise Training in Non-Small Cell Lung Cancer
Brief Title: Pre Radiotherapy Daily Exercise Training in Non-Small Cell Lung Cancer
Acronym: PRIME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Morten Quist, Principal Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: JRTE; H-16048479 (Other Grant/Funding Number: Toyota Foundation)
Record Dates: First submitted 2017-02-08; First posted 2017-02-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2022-10

CONDITIONS: Non-Small Cell Lung Cancer Stage; Chemoradiation
Keywords: Aerobic exercise; Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise + usual care (Experimental): The supervised exercise training is carried out on a ergometer cycle as individual daily (mon-fri) training and each exercise training session consists of 20min.
  The training comprised a warm-up phase followed by 3 exercise phases. Warm-up consisted of 5min light stationary cycling, adjusted to 50-60% of the patients peak power output determine at the incremental cycle test (iPPO). The first exercise phase comprised of 5min interval training consisting of 5x30 sec intervals at 80-95% of the patient's iPPO. Between each interval, there is a 30 sec pause. The 2nd exercise phase consisted of 5min continuous cycling at an intensity equaling 80% of the patient's iPPO. The 3rd exercise phase was similar to the first exercise phase. Intensities increased progressively from the first week to the last week (from 50%, 80% and 70% of iPPO according to the three different phases to 60%, 95% and 80 % of iPPO respectively.
  Interventions: Other: Exercise +
- Control - usual care (Experimental): The patients randomized to the control group received no training but will be wearing the activity tracker during the intervention.
  Interventions: Other: Control +

INTERVENTIONS:
Other: Exercise + — Usual care
  Arms: Exercise + usual care
Other: Control + — Usual care
  Arms: Control - usual care

SUMMARY:
The aim of this study is to evaluate the feasibility and the effect of daily, individual, supervised and structured exercise training before radiotherapy in patients diagnosed with Non-Small Cell Lung Cancer. Primary outcome is maximal oxygen uptake (VO2peak). The hypotheses are that patients who undergo daily exercise training will increase VO2peak, functional capacity (measured by 6-minute walk test (6MWD)) and lung function (forced expired volume in one second (FEV1)).

DETAILED DESCRIPTION:
Pre intervention screening: Each patient was screened by a clinical nurse specialist prior to participating in the study. Before baseline and post test the patient was screened by a research physiotherapist and/or human physiology students. If one of the following criteria were met, the patient was prohibited from being tested on that day: diastolic blood pressure <45 or >95, heart rate (HR) at rest >115/min, temperature > 38 0C, respiratory rate at rest >30/min, infection requiring treatment, fresh bleeding, total leucocyte count <1.0 109/L or platelets <50 109/L.

Control - Usual care: The patients randomized to the control group received no training but conducted baseline and post test (6MWD, spirometry, VO2peak and questionnaires) just as the intervention group. Furthermore, patients in control were equipped with a Garmin vivo-smart HR® activity tracker every day in 24h during the course of radiotherapy treatment.

Intervention - The patients randomized to the intervention group received daily training and conducted baseline and post test (6MWD, spirometry, VO2peak and questionnaires). Furthermore, patients were equipped with a Garmin vivo-smart HR® activity tracker every day in 24h during the course of radiotherapy treatment.

The supervised daily training was carried out individually and each session had a duration of 20 minutes before patients individual prescribed radiotherapy. Training was conducted at National Hospital of Denmark: Department of Radiation Oncology , section 3981, entry 39. supervised by a research physiotherapist and/or human physiology students.

Statistical analysis sample size: According to the sample size the calculation is performed on the basis of alteration in VO2peak from the study "EXHALE" (55 patients who completed a 6 weeks training period). The calculation is based on an increase of 200 ml/min in VO2peak for patients in the intervention group (SD = 2,48) and it is assumed that the patients in the control group will have a reduction of 100 ml/min (SD = 2,48). Assumptions for calculation of patient numbers are as follows: Type 1 error 0.05, type 2 error 0.20, SD 2.48.

This leads to a total number of 24 patients (12 in each arm). A drop-out rate of 40% is included. Therefore another 16 patients is added, which gives a sample size of 40 patients (20 in each arm).

Data entry is carried out in the Open Clinica and data analyses will be performed using the computer programs R-Studio/R and SPSS. Data from questionnaires will be analyzed by SPSS. All other data will be analyzed by R.

Differences between groups will be analyzed by an unparried t-test whereas differences within groups will be analyzed by a parried t-test. All categorical data are analyzed using the Pearson χ2 tests. Other data (e.g., from questionnaires) are analyzed using logistic regression and chi square or Mantel Haenzel test. Significance level is set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NSCLC who are treated with concomitant chemo- and radiotherapy.
* Age: > 18 year
* WHO performance status 0-1

Exclusion Criteria:

* Patients with any symptoms or circumstances that advise against physical activity.
* Symptomatic heart disease e.g. arrhythmia or myocardial infarction within the last three months.
* Congestive heart failure
* Patients who do not read and speak Danish.
* Brain or bone metastases;
* Prolonged bone marrow suppression
* Anti-coagulant treatment
* Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-04-03 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum oxygen uptake - VO2peak | Change from baseline at 7 weeks
  The primary outcome will be VO2peak, assessed with an aerobic capacity (VO2peak) incremental cycle ergometer test performed on a Monark ergometer 839E cycle.
  At baseline, human physiology students will carry out the incremental cycle test. A physiotherapist who is blinded to the groups wherein the patients are allocated will carry out the posttest.
  The test consist of a warm-up phase at 10-50 w. After warm-up the load increases by 5-10 w every 60 sec until exhaustion or a possible symptom limitation (e.g. dizziness, sudden pain, vomiting sensation). To analyze the expired gases patients are going to wear a Hans Rudolf Mask during the test. Expired gases will be analyzed continuously by a metabolic breath-by-breath analysis and calculated as an average over 15 sec using the Oxycon Pro. Jaeger measurement system.

SECONDARY OUTCOMES:
Functional capacity | Baseline and 7 weeks
  Functional capacity is measured by a 6 MWD test. The test is carried out over a pre-measured distance of 20 meters, in compliance with the American Thoracic Society (ATS) statement. After the test the patients will rate the breathing on Borg Scale for dyspnea.
Forced Expiratory Volume in one second | Baseline and 7 weeks
  Forced Expiratory Volume in 1 second (FEV1) is measured using a standard spirometry in a standing position with the use of the Oxycon Pro, Jaeger measurement system.
Lung Function | Baseline and 7 weeks
  Ventilation (VE), Breath frekvens (BF) and tidal volume (Vt) measured by indirect calorimetry.
Hypoxia in tumor | Baseline and 7 weeks
  The extent of hypoxia in human tumors assessed by dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI).
Stroke volumen | Baseline, selected test samples during training intervention and 7 weeks
  Stroke volumen will be measured by a ClearSight System
Cardiac output | Baseline, selected test samples during training intervention and 7 weeks
  Cardiac output will be measured by a ClearSight System
Systemic vascular resistance | Baseline, selected test samples during training intervention and 7 weeks
  Systemic vascular resistance (SVR) will be measured by a ClearSight System
Safety: Sports-injury, Pain, Neuropathies, Nausea/vomiting, Fatigue etc. | Baseline, during intervention and 7 weeks
  Serious adverse events and adverse events (e.g.)sports-injury, pain, neuropathies, nausea/vomiting, fatigue, neutropenia, fever, diarrhoea, hospitalisation and infection
Respiratory exchange ratio (RER) | Change from baseline at 7 weeks
  To analyze the expired gases patients are going to wear a Hans Rudolf Mask during a incremental cycle ergometer test. Expired gases will be analyzed continuously by a metabolic breath-by-breath analysis and calculated as an average over 15 seconds using the Oxycon Pro. Jaeger measurement system.
Rated Perceived Exertion (RPE) Scale | Change from baseline at 7 weeks
  In the final seconds of the incremental cycle ergometer test self-perceived exertion perception and dyspnoea will be noted.

OTHER OUTCOMES:
Overall survival rate | 26 weeks and 52 weeks
  Overall survival be measured from inclusion until death or 26 weeks or 52 weeks
Physical Activity | Change from baseline at 7 weeks
  Physical Activity - International Physical Activity Questionnaire Long (IPAQ-L).
Quality of life and wellbeing | Change from baseline at 7 weeks
  Quality of life and wellbeing - Functional Assessment of Cancer Therapy - Lung (FACT-L).
Anxiety and depression | Change from baseline at 7 weeks
  Anxiety and depression - Hospital Anxiety and Depression Scale (HAD)
Activity Data | Every day in 24h during the course of radiotherapy treatment
  Steps, distance and intensity minutes measured by Garmin vivo-smart HR® activity tracker.

CONTACTS AND LOCATIONS:
Overall Officials: Morten Quist, Post. doc, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- University Hospital of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No